CLINICAL TRIAL: NCT05643521
Title: The Acute Effects of Eucaloric and Hypocaloric Carbohydrate Restriction on Liver Fat Content and Metabolism in Obese Individuals
Acronym: FixedCarb
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other); Nutrition Exercise and sports Copenhagen University (Unknown)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, Principal investigator, MD, PhD Affiliation: Hvidovre University Hospital, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: FixedCarb - H-22035189
Record Dates: First submitted 2022-11-22; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: NAFLD; Overweight and Obesity; Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Overweight; Obesity; Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Randomized diet intervention study in a cross over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Experimental): 2 days of eucaloric control diet prior to MRS estimating liver fat (control arm)
  Interventions: Other: Dietary composition of macronutrients and calories
- Hypocaloric low carbohydrate (Experimental): 2 days of eucaloric control diet + 2 days of hypocaloric (500-600 kcal m/f) low carbohydrate diet prior to liver fat estimated by MRS and metabolic testday.
  Interventions: Other: Dietary composition of macronutrients and calories
- Eucaloric low carbohydrate (Experimental): 2 days of eucaloric control diet + 2 days of eucaloric low carbohydrate diet prior to liver fat estimated by MRS and metabolic testday.
  Interventions: Other: Dietary composition of macronutrients and calories

INTERVENTIONS:
Other: Dietary composition of macronutrients and calories — Carbohydrate restriction

SUMMARY:
The primary aim of this study is to investigate the acute changes in liver fat content in response to a fixed carbohydrate restriction (i.e. intake of 60g/day or 70g/day for women and men, respectively) in individuals with obesity. This will be performed both as 2 days of very low calorie diet (500 and 600 kcal/day for women and men, respectively) and 2 days of eucaloric low carbohydrate diet.

ELIGIBILITY:
Inclusion Criteria:

* Men (30-75 years) and postmenopausal women 45-75 years old
* Hba1c <48 mmol/mol without antidiabetic treatment
* Obese (BMI 27-40 kg/m2)
* Non smokers

Exclusion Criteria:

* Anemia (hemoglobin <8 mmol/L for men and <7 mmol/L for women)
* TSH outside reference range
* Medication known to influence glucose metabolism or appetite regulation
* Contraindications for MR-scan: abdominal height exceed limitations of the MR-scanner, pacemaker or other electronic device implanted, implanted metal devices, severe claustrophobia
* Food allergies (including lactose and gluten intolerance), vegetarian/vegan diet or following specific dietary plans
* Alcohol consumptions >84/168 g/week (women/men)
* Strenuous activity level > 120 minutes per week
* >5 kg weight loss within the last three months or previous bariatric surgery
* High risk of fibrosis of the liver (estimated by FIB4 score > 3,25)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the 1H-Magnetic Resonance Spectroscopy (MRS) determined liver TG content. | After 2 days completion of dietary intervention
  We will compare MRS of liver TG after each of the two interventions (2 days of VLCD or 2 days of LC) with MRS liver TG obtained after 2 days of eucaloric conventional diet.

SECONDARY OUTCOMES:
Secondary outcomes are fasting and postprandial plasma glucose, insulin, and plasma TG concentrations after 2 days VLCD or LC compared with 2 days of eucaloric conventional diet. | After 2 days completion of dietary intervention

OTHER OUTCOMES:
Explorative outcomes | After 2 days completion of dietary intervention
  Explorative outcomes are the effects of VLCD and LC on subsequent food intake in response to an ad libitum lunch meal.